CLINICAL TRIAL: NCT01408914
Title: Randomized Trial of High-Dose Rifampin in Patients With New, Smear-Positive TB
Brief Title: Trial of High-Dose Rifampin in Patients With TB
Acronym: HIRIF
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Harvard University Faculty of Medicine (Other)
Collaborators: National Institute of Allergy and Infectious Diseases (NIAID) (NIH); Sanofi (Industry); Harvard School of Public Health (HSPH) (Other); Brigham and Women's Hospital (Other); University of Liverpool (Other); St George's, University of London (Other); University of Florida (Other); Socios en Salud (Unknown)
Responsible Party: Principal Investigator, Carole Mitnick, Associate Professor, Harvard University Faculty of Medicine
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 11-0050; 5U01AI091429-03 (NIH)
Record Dates: First submitted 2011-08-02; First posted 2011-08-03 (Estimated); Results first posted 2017-07-13 (Actual); Last update posted 2017-11-20 (Actual); Status verified 2017-10

CONDITIONS: Tuberculosis
MeSH Terms: conditions — Tuberculosis | interventions — Rifampin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- RIF 600 (No Intervention)
- RIF 900 (Experimental)
  Interventions: Drug: Higher-Dose Rifampin
- RIF 1200 (Experimental)
  Interventions: Drug: Higher-Dose Rifampin

INTERVENTIONS:
Drug: Higher-Dose Rifampin — The intervention phase of this trial will last 8 weeks. During that time, subjects will receive the following companion drugs: isoniazid (INH, 5 mg/kg/day), ethambutol (EMB, 20 mg/kg/day), and pyrazinamide (PZA, 25 mg/kg/day), pyridoxine (50 mg), the standard doses used in treatment. Subjects will also be randomized to receive one of the following weight-based doses of the study drug, rifampin (RIF): 10 mg/kg/day (standard dose, control), 15 mg/kg/day (intervention 1), 20 mg/kg/day (intervention 2). All patients will receive at least standard dose of RIF, the efficacy of which in multidrug-treatment for TB is well established. Placebo will be used to control only the additional RIF capsules provided in the intervention arms.
  Other Names: rifadin, rifampicin
  Arms: RIF 1200; RIF 900

SUMMARY:
The purpose of this study is to evaluate the potential of high doses of rifampin (RIF) to shorten treatment for tuberculosis (TB) without causing more adverse events. The hypotheses are that higher doses of RIF will result in higher blood concentrations of RIF; higher blood concentrations will result in tuberculosis bugs being killed more quickly; and, both of these will happen without more adverse events. Patients with active, infectious, drug-susceptible TB who agree to participate will be randomly assigned to 1 of 3 doses of RIF. All patients will also receive standard doses of regular (3) companion drugs for 2 months of daily, supervised therapy. The study will assess the following among the 3 study arms (oral doses of RIF 10, 15 & 20 mg/kg/day) during the initial 8 weeks of treatment: 1) the amount of RIF in the blood after at least 14 days of treatment; 2) the difference in the number of tuberculosis bugs killed; 3) the frequency of adverse events.

DETAILED DESCRIPTION:
This is a Phase II, multi-site, dose-ranging trial comparing 3 doses of RIF in a multidrug regimen for treatment of smear-positive, pulmonary TB. The intervention phase of this prospective, randomized, double-blinded trial will last 8 weeks, the duration of the standard "intensive" phase for short-course chemotherapy for TB. During that time, subjects will receive the following companion drugs: isoniazid (INH, 5 mg/kg/day), ethambutol (EMB, 20 mg/kg/day), and pyrazinamide (PZA, 25 mg/kg/day), pyridoxine (50 mg), the standard doses used in treatment. Subjects will also be randomized to receive one of the following weight-based doses of the study drug, rifampin (RIF): 10 mg/kg/day (standard dose, control), 15 mg/kg/day (intervention 1), 20 mg/kg/day (intervention 2). All patients will receive at least standard dose of RIF, the efficacy of which in multidrug-treatment for TB is well established. Placebo will be used to control only the additional RIF capsules provided in the intervention arms. Subjects, clinicians, and laboratory staff will be blinded to study arm. All patients in the same weight band will receive the same total number of tablets (fixed-dose combination plus RIF and/or placebo). Blinding is essential to reduce the probability of biased reporting of adverse events.

After randomization, other covariates that may result in heterogeneity within strata (e.g., presence of cavitation, HIV serostatus), will be adjusted for in analyses. It is important to maintain the ability to measure the effect (if any) of these potential characteristics on treatment outcome. If we were to stratify on these characteristics, we could not estimate their confounding (or interaction) effect. All doses will be delivered orally and fully supervised. All patients will receive weight-based doses of fixed-dose combinations according to package inserts. This will be supplemented by active RIF capsules or placebos, or both, according to weight and treatment arm. They will also all receive 50 mg of pyridoxine to prevent peripheral neuropathy, a common side effect of INH.

ELIGIBILITY:
Inclusion Criteria:

* Newly diagnosed pulmonary TB with acid-fast bacilli (>=2+) in a stained sputum smear, ultimately confirmed by culture.
* Susceptibility of isolate to INH and RIF by HAIN test.
* Willingness to undergo HIV testing according to the National Health Guidelines for TB control in Peru. The study will also consider patients who have had negative HIV serostatus documented within six months prior to enrollment or if verifiable positive serostatus was documented using a validated test any time previously.
* Age >/= 18 years and <61 years.
* Signed informed consent.
* Negative serum pregnancy test (women of childbearing potential).
* Women with child-bearing potential must agree to practice a double-barrier method of birth control during treatment. Adequate contraceptives (condoms and spermicide) will be provided by the study to avoid pregnancy among female subjects.
* Karnofsky score of at least 50 (requires considerable assistance and frequent medical care).
* Intends to remain in jurisdiction of health center during study and follow up.

Exclusion Criteria:

* Body weight <30 kg.
* Prior treatment with multidrug anti-TB therapy for more than one month.
* Resistance on HAIN to INH and/or RIF. These patients will be treated according to local programmatic guidelines.
* Central nervous system or miliary TB.
* Clinical or radiological signs suggestive of pericardial or pleural involvement.
* Presence of significant hemoptysis. Patients who cough up frank blood (more than blood-streaked sputum) will not be eligible for enrollment.
* Known intolerance to any of the study drugs; use of concomitant drugs that interfere with the pharmacokinetics of anti-TB drugs; use of concomitant hepatotoxic drugs (other than companion study drugs) for which potential drug interactions or synergistic toxicity are known: boosted protease inhibitors, non-nucleoside reverse transcriptase inhibitors, azole antifungals and statins; use of antibiotics that are contraindicated during the study's TB therapy; current daily use of acetaminophen or paracetamol for two weeks or more.
* History of liver disease.
* Uncontrolled condition that might interfere with drug absorption, distribution, metabolism or excretion (i.e. chronic gastrointestinal disease, renal insufficiency defined by creatinine clearance <60mL/min).
* Uncontrolled diabetes mellitus (HbA1c>7.5%).
* Refusal to be tested for HIV infection; HIV infection with contraindication for treatment with efavirenz (including resistance).
* Pulmonary silicosis.
* Breastfeeding.
* Rifampin contraindications such as hypersensitivity or jaundice.
* Likely difficulty adhering to the protocol, as assessed by the investigator.
* Laboratory results in the 14 days preceding enrollment showing:

  1. Serum amino alanine transferase (ALT) >2 times upper limit of normal
  2. Serum total bilirubin concentration >2.5 times upper limit of normal
  3. Serum creatinine concentration > 2 times upper limit of normal and/or creatinine clearance <60 mL/min
  4. Hemoglobin concentration < 7.0 g/dL
  5. Platelet count < 150,000/mm3
  6. White blood count <4500 cells/μL.
* Having a serological test positive for HBVsAg (hepatitis B virus surface antigen) or for HCVAb (hepatitis C virus antibody)test.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 180 (Actual)
Dates: Start 2013-09; Primary Completion 2016-04 (Actual); Study Completion 2016-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Carole D Mitnick, Sc.D, Principal Investigator — Harvard Medical School (HMS and HSDM); Geraint Davies, B.M., Ph.D, Principal Investigator — University of Liverpool
Locations (4):
- University of Florida, Gainesville, Florida, United States
- Socios En Salud Sucursal Perú, Lima, Peru
- United Kingdom (2):
  - School of Clinical Sciences at University of Liverpool, Liverpool
  - St. George's University of London, London

REFERENCES:
- [Background] Milstein M, Lecca L, Peloquin C, Mitchison D, Seung K, Pagano M, Coleman D, Osso E, Coit J, Vargas Vasquez DE, Sanchez Garavito E, Calderon R, Contreras C, Davies G, Mitnick CD. Evaluation of high-dose rifampin in patients with new, smear-positive tuberculosis (HIRIF): study protocol for a randomized controlled trial. BMC Infect Dis. 2016 Aug 27;16(1):453. doi: 10.1186/s12879-016-1790-x. PMID 27567500
- [Result] Peloquin CA, Velasquez GE, Lecca L, Calderon RI, Coit J, Milstein M, Osso E, Jimenez J, Tintaya K, Sanchez Garavito E, Vargas Vasquez D, Mitnick CD, Davies G. Pharmacokinetic Evidence from the HIRIF Trial To Support Increased Doses of Rifampin for Tuberculosis. Antimicrob Agents Chemother. 2017 Jul 25;61(8):e00038-17. doi: 10.1128/AAC.00038-17. Print 2017 Aug. PMID 28559269
- [Derived] Mackay E, Platt G, Peloquin CA, Brooks MB, Coit JM, Velasquez GE, Pertinez H, Vargas D, Sanchez E, Calderon RI, Jimenez J, Tintaya K, Garcia D, Osso E, Lecca L, Mitnick C, Davies GR. Impact of Pharmacogenetics on Pharmacokinetics of First-Line Antituberculosis Drugs in the HIRIF Trial. J Infect Dis. 2025 Aug 14;232(2):e258-e265. doi: 10.1093/infdis/jiaf195. PMID 40239986

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment was done through routine passive case detection in operation at ambulatory facilities in the Peruvian public health system (DISA IV-Lima Este and DISA V- Lima Ciudad).
Pre-assignment Details: 180 participants were randomized in a 1:1:1 allocation to the 10, 15, and 20 mg/kg treatment arms.
Groups:
- 10 mg/kg: 10 mg/kg RIF
- 15 mg/kg: 15 mg/kg RIF
- 20 mg/kg: 20 mg/kg RIF
Period: Overall Study
Arm/Group | 10 mg/kg | 15 mg/kg | 20 mg/kg
Started | 60 | 60 | 60
Completed | 48 | 48 | 47
Not Completed | 12 | 12 | 13
Not completed — Could not complete tx in protocol period | 5 | 5 | 6
Not completed — Lost to Follow-up | 4 | 1 | 2
Not completed — Physician Decision | 1 | 1 | 0
Not completed — Withdrawal by Subject | 1 | 0 | 1
Not completed — Moved out of study jurisdiction | 1 | 1 | 0
Not completed — Late exclusion | 0 | 3 | 3
Not completed — Change in local TB/HIV norms | 0 | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | 10 mg/kg | 15 mg/kg | 20 mg/kg | Total
Number analyzed (Participants) | 60 | 60 | 60 | 180
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 24 [21 to 37] | 25 [20 to 35] | 27 [22 to 37] | 25 [21 to 37]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 21 | 19 | 26 | 66
  Male | 39 | 41 | 34 | 114
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 60 | 60 | 59 | 179
  Not Hispanic or Latino | 0 | 0 | 1 | 1
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 1 | 1 | 3
  Asian | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0
  White | 0 | 2 | 1 | 3
  More than one race | 57 | 51 | 54 | 162
  Unknown or Not Reported | 2 | 6 | 4 | 12

OUTCOME MEASURES:

1. Primary Outcome: Steady State Pharmacokinetic Exposure of RIF
Description: The endpoint is the (dimensionless) ratio of AUC0-6 mcg/ml*h to MIC99.9 mcg/ml
Time Frame: At any time during the intensive phase of treatment, after steady state has been reached (at a minimum, after 14 days of daily RIF delivery)
Population: Analysis was completed in 168 participants evaluable for pharmacokinetics, as samples were unable to be collected in 12 study participants.
Measure: Median (Inter-Quartile Range); unit: Ratio
Arm/Group | 10 mg/kg | 15 mg/kg | 20 mg/kg
Number analyzed (Participants) | 58 | 57 | 53
Ratio | 115.6988 [59.1233 to 197.5544] | 201.9725 [144.1413 to 460.2869] | 284.4278 [175.2923 to 399.2127]

2. Secondary Outcome: Sputum Culture Sterilization During the Initial 8 Weeks of Treatment
Description: Number of participants that are sputum culture (in LJ) negative for TB at 8 weeks
Time Frame: Until 8 weeks of treatment are completed
Measure: Count of Participants; unit: Participants
Arm/Group | 10 mg/kg | 15 mg/kg | 20 mg/kg
Number analyzed (Participants) | 60 | 60 | 60
Participants | 46 | 44 | 45

3. Secondary Outcome: Incidence of Rifampin-related Grade 2 or Higher Adverse Events
Description: Number of participants experiencing at least one rifampin-related grade 2 or higher adverse events during the initial 8 weeks of treatment and up to four weeks after.
Time Frame: Throughout the 12 weeks post treatment initiation
Measure: Count of Participants; unit: Participants
Arm/Group | 10 mg/kg | 15 mg/kg | 20 mg/kg
Number analyzed (Participants) | 60 | 60 | 60
Participants | 26 | 31 | 23

ADVERSE EVENTS:
Arm/Group | 10 mg/kg | 15 mg/kg | 20 mg/kg
Serious Adverse Events (participants affected / at risk) | 2/60 | 1/60 | 5/60
Other Adverse Events (participants affected / at risk) | 26/60 | 30/60 | 21/60
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 10 mg/kg (N=60) | 15 mg/kg (N=60) | 20 mg/kg (N=60)
Respiratory (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 2 (2)
Hepatic (Hepatobiliary disorders) | 1 (1) | 1 (1) | 2 (2)
Neurological (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 1 (1)
OB-GYN (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 10 mg/kg (N=60) | 15 mg/kg (N=60) | 20 mg/kg (N=60)
Blood and lymphatic system disorders (Blood and lymphatic system disorders) | 1 (1) | 1 (1) | 1 (1)
Gastrointestinal disorders (Gastrointestinal disorders) | 4 (4) | 13 (15) | 4 (5)
Hepatobiliary disorders (Hepatobiliary disorders) | 16 (16) | 13 (13) | 12 (12)
Immune system disorders (Immune system disorders) | 0 (0) | 0 (0) | 1 (1)
Investigations (Investigations) | 1 (1) | 1 (1) | 0 (0)
Metabolism and Nutrition Disorders (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0)
Musculoskeletal and connective tissue disorders (Musculoskeletal and connective tissue disorders) | 2 (2) | 3 (3) | 3 (3)
Nervous system disorder (Nervous system disorders) | 1 (1) | 1 (1) | 0 (0)
Respiratory, thoracic and mediastinal disorders (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 3 (3) | 1 (1)
Skin and subcutaneous tissue disorders (Skin and subcutaneous tissue disorders) | 6 (6) | 1 (1) | 7 (8)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No